CLINICAL TRIAL: NCT06113978
Title: Fifteen Years' Experience of Thoracoscopic Sympathetic Chain Interruption for Palmar Hyperhidrosis in Children and Adolescents; Evaluation of Different Techniques
Brief Title: Thoracoscopic Sympathetic Chain Interruption for Palmar Hyperhidrosis in Patients Below 18
Acronym: MISforPPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Muhammad Abdelhafez Mahmoud, MD (Other)
Responsible Party: Sponsor-Investigator, dr. Muhammad Abdelhafez Mahmoud, MD, Lecturer of pediatric surgery, Al-Azhar Faculty of Medicine, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlAzharThoracoscSympathforPPH
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Hyperhidrosis; Children, Adolescents; Thoracoscopic Sympathetic Chain Interruption; Sympathetic Disorder
Keywords: Palmar hyperhidrosis;; Thoracoscopic sympathectomy;; Compensatory sweating;; Pediatrics,; Adolescents
MeSH Terms: conditions — Hyperhidrosis; Autonomic Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: This retrospective study was conducted at the Department of pediatric surgery, Al-Azhar University Hospitals in the period from April 2008 to March 2023, involving patients of both sexes, below 18 years of age, suffering from severe bothersome bilateral palmar hyperhidrosis, managed by thoracoscopic bilateral simultaneous sympathetic chain interruption.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracoscopic sympathectomy for palmar hyperhidrosis in children and adolescents (Active Comparator): Medical file records of patients of both sexes, below 18 years of age, suffering from significant bilateral palmar hyperhidrosis, managed by thoracoscopic bilateral simultaneous sympathectomy.
  Interventions: Procedure: Thoracoscopic sympathectomy
- Thoracoscopic sympathotomy for palmar hyperhidrosis in children and adolescents (Active Comparator): Medical file records of patients of both sexes, below 18 years of age, suffering from significant bilateral palmar hyperhidrosis, who underwent thoracoscopic bilateral simultaneous sympathotomy.
  Interventions: Procedure: Thoracoscopic sympathotomy
- Thoracoscopic sympathetic chain clipping for palmar hyperhidrosis in children and adolescents (Active Comparator): Medical file records of patients of both sexes, below 18 years of age, suffering from significant bilateral palmar hyperhidrosis, treated by thoracoscopic bilateral simultaneous sympathetic chain clipping.
  Interventions: Procedure: Thoracoscopic sympathetic chain clipping

INTERVENTIONS:
Procedure: Thoracoscopic sympathectomy — Medical file records of patients of both sexes, below 18 years of age, suffering from significant bilateral palmar hyperhidrosis, managed by thoracoscopic bilateral simultaneous sympathectomy.
  Arms: Thoracoscopic sympathectomy for palmar hyperhidrosis in children and adolescents
Procedure: Thoracoscopic sympathotomy — Medical file records of patients of both sexes, below 18 years of age, suffering from significant bilateral palmar hyperhidrosis, who underwent thoracoscopic bilateral simultaneous sympathotomy.
  Arms: Thoracoscopic sympathotomy for palmar hyperhidrosis in children and adolescents
Procedure: Thoracoscopic sympathetic chain clipping — Medical file records of patients of both sexes, below 18 years of age, suffering from significant bilateral palmar hyperhidrosis, treated by thoracoscopic bilateral simultaneous sympathetic chain clipping.
  Arms: Thoracoscopic sympathetic chain clipping for palmar hyperhidrosis in children and adolescents

SUMMARY:
In this study, the investigators aim to present fifteen years' experience of thoracoscopic sympathetic chain interruption for primary palmar hyperhidrosis in children and adolescents; evaluation of 3 different techniques (sympathectomy, sympathotomy, and clipping) regarding demographic data, surgical outcomes, complications, compensatory sweating, and patients' satisfaction.

DETAILED DESCRIPTION:
Primary palmar hyperhidrosis (PPH) is a severely devastating autonomic disorder that can affect any patient regardless age, even pediatrics. Thoracoscopic sympathetic chain interruption offers a definitive effective therapy. In this study, the investigators aim to assess the outcomes of thoracoscopic management of palmar hyperhidrosis in a large cohort of children younger than 18 years old with severe PPH, using sympathetic chain interruption either by sympathectomy, sympathotomy or clipping, to provide a methodology focused on the long-term outcomes of those procedures.

Patients and Methods: This is a retrospective study that included all children who underwent thoracoscopic sympathectomy, sympathotomy, or clipping for severe PPH, from April 2008 to March 2023 were assessed retrospectively. Demographic data, postoperative outcome, complications, compensatory sweating and satisfaction were analyzed.

Surgical procedures:

General anesthesia was used, with an ordinary endotracheal tube, by an experienced anesthesiologist who used one lung ventilation anesthesia to control the patient's O2-enriched ventilation in a low-volume/high-frequency technique, with alternating brief periods of apnea. The patient was placed in the semi-Fowler position, which is the dorsal decubitus position with the arms abducted and fixed at 90 degrees. The trunk was elevated by 30-40 degrees; as elevation helped displace the lungs downwards. A slight bed elevation at the knee level was useful to safely place the patients and prevent them from slipping down during the procedure.

To access the thoracic cavity, the investigators used the two-port video thoracoscopy using two 5 mm ports via 2 mini-incisions. The camera (30º scope) port was placed laterally at the fourth or fifth intercostal space (depending on the age of the patient) just posterior to the anterior axillary fold created by the pectoralis major muscle. The second port (for electrocautery instrument (hook) was laterally inserted in the third/fourth intercostal space at the mid-axillary line as that approach provides excellent aesthetic results. A CO2 pneumothorax pressure of 5-8 mmHg was used according to patient's age and body built. The posterior parietal pleura was incised just lateral to neck of 3rd rib and further dissected down to identify the thoracic sympathetic chain.

A-Thoracoscopic sympathectomy: A segment of the thoracic sympathetic chain at the intended levels is resected using hook electrothermoablation.

B-Thoracoscopic sympathotomy technique (VATS): The sympathetic chain is just cut at the desired levels without excision.

C-Thoracoscopic clipping technique: Titanium clips are applied on the desired level without cutting. Then, after completion of the procedure, CO2 pneumothorax was deflated, permitting full lung inflation under vision, without need for chest tube placement, ports removal, and port-sites closure by absorbable sutures with full awake recovery from anesthesia. Post operative routine chest x-ray was done to detect any residual pneumothorax and to assess the location of clips in clipping group.

Statistical Analysis:

Data were collected, revised, coded, and entered to the Statistical Package for Social Science (SPSS), IBM, version 23. The qualitative data were presented as numbers and percentages, while the quantitative data were presented as means, standard deviations, and ranges when their distribution was found to be parametric. Independent t-test and Chi-square tests were used to compare both groups. The p-value was considered significant if < 0.05.

Discussion: will explore the different treatment modalities for PPH in children and adolescents, mentioning the medical/conservative methods, then focusing on the surgical option, that is thoracoscopic sympathetic chain interruption, either by sympathectomy, sympathotomy, and clipping for almost permanent remedy of PPH in pediatric age group younger than 18 years old. Points of discussion will include demographic data, follow-up period, surgical outcomes and complications, compensatory sweating, and patients' satisfaction.. The results obtained will be compared among the 3 groups and also compared to the previously published articles.

Finally, the investigators will conclude whether or not there is a better technique among the 3 modalities that gives the best durable outcome with the least complications.

ELIGIBILITY:
Inclusion Criteria:

* visible exaggerated bilateral symmetrical sweating with impaired daily activities (such as shaking hands, writing and drawing),
* without other apparent cause (e.g., hyperthyroidism, DM, or TB).

Exclusion Criteria:

* secondary hyperhidrosis,
* nocturnal sweating,
* recurrent cases, and
* patients older than 18 years

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
success rate | 2 years
  number of patients with post operative dry hands
compensatory sweating | 2 years
  number of patients with post operative compensatory sweating
patient satisfaction rate | 2 years
  number of patients simply questioned for outcome satisfaction (either very satisfied, satisfied, or dissatisfied)

SECONDARY OUTCOMES:
complications | 2 years
  number of complications
recurrence rate | 2 years
  number of recurrent cases

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmed A Alzayyat, MD, Study Director — Deputy Dean, professor, Pediatric Surgery Department, Al-Azhar University
Locations (1):
- Pediatric Surgery Department, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author but could not be sent owing to the medicolegal aspect of the hospital policy.
Supporting Information: Study Protocol, CSR
Time Frame: from today indefinitely
Access Criteria: for other colleagues who may be interested with the study topic
URL: http://orcid.org/0000-0002-6328-6419

REFERENCES:
- Available data/document: Study Protocol: orcid.org/0000-0002-6328-6419 — http://orcid.org/0000-0002-6328-6419 — the corresponding author (sponsor/principal investigator) of this work can be contacted for help anytime by colleagues who concern